CLINICAL TRIAL: NCT01469169
Title: A Multi-center, Non-randomized, Open Label, Single-arm Study to Evaluate the Efficacy, Safety, and Pharmacokinetics (PK) of BAY q 6256 (Iloprost) Inhalation in Patients With Pulmonary Arterial Hypertension (PAH)
Brief Title: Inhaled Iloprost (Ventavis): Efficacy, Safety, and Pharmacokinetics (PK) Confirmation Study
Acronym: IBUKI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15503
Record Dates: First submitted 2011-11-08; First posted 2011-11-10 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Hypertension, Pulmonary
Keywords: Iloprost; Inhalation; Pulmonary Hypertension; Pulmonary Artery Hypertension; Japanese Patients
MeSH Terms: conditions — Hypertension, Pulmonary; Respiratory Aspiration; Familial Primary Pulmonary Hypertension | interventions — Iloprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Iloprost (Ventavis inhaled, BAYQ6256)

INTERVENTIONS:
Drug: Iloprost (Ventavis inhaled, BAYQ6256) — 2.5 μg or 5.0 μg BAYQ6256 per inhalation session (Inhalation session is to be conducted 6 to 9 times per day with dosing intervals of at least 2 hours.)

SUMMARY:
This study is to investigate the efficacy, safety, and Pharmacokinetics (PK) of Inhaled Iloprost (Ventavis) therapy in Japanese pulmonary arterial hypertension (PAH) patients in Main Treatment Phase (12 weeks) and to investigate the safety, tolerability, and efficacy of longterm Inhaled Iloprost (Ventavis) therapy in Japanese PAH patients in Extension Phase.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 to 75 years
* Symptomatic Pulmonary Artery Hypertension (PAH) classified (Dana Point Classification 1)
* New York Heart Association (NYHA)/World Health Organization (WHO) functional class III or IV
* PAPmean at rest > 25 mm Hg, Pulmonary capillary wedge pressure (PCWP) or left ventricular end-diastolic pressure </= 15 mm Hg and Pulmonary Vascular resistance (PVR) >/= 240 dyn.sec.cm-5 (>/= 400 dyn.sec.cm-5 for patients treated with both endothelin receptor antagonist (ERA) and phosphodiesterase-5 inhibitor (PDE5i) ) as measured by Right Heart Catheter test
* Women of childbearing potential and men must agree to use adequate contraception when sexually active

Exclusion Criteria:

* Baseline 6-minute walk distance of less than 100 meters or more than 500 meters
* Subjects with critical severe PAH
* Forced Expiratory Volume in 1 second (FEV1)/Forced Vital Capacity (FVC) ratio < 60% and/or Total Lung Capacity (TLC) < 70% predicted (especially at interstitial lung disease, TLC < 60% predicted)
* Clinically relevant obstructive lung disease (e.g. asthma or chronic obstructive pulmonary disease )
* More than mild patchy interstitial lung disease on High Resolution Computerized Tomography (HRCT)
* History of left-sided heart disease
* Uncontrolled systemic hypertension as evidenced by systolic blood pressure >/= 160 mm Hg or diastolic blood pressure >/= 100 mm Hg on repeated measurement
* Systemic hypotension with systolic blood pressure < 85 mm Hg

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-06-19 (Actual); Primary Completion 2014-12-26 (Actual); Study Completion 2016-12-14 (Actual)

PRIMARY OUTCOMES:
Change in Pulmonary vascular resistance (PVR) from screening (baseline) to week 12 (after inhalation) | At baseline and 12 weeks
Number of participants with adverse events as a measure of safety and tolerability | Up to 52 weeks
Area under the plasma concentration vs time curve from start of inhalation to infinity after single inhalation (AUC) | At baseline, 12 weeks, 52 weeks and over 52 weeks
Maximum drug concentration in plasma after start of inhalation (Cmax) | Up to 12 weeks
Number of participants with adverse events as a measure of safety and tolerability | Over 52 weeks

SECONDARY OUTCOMES:
Change of Pulmonary vascular resistance index (PVRI) from baseline to week 12 | At baseline and 12 weeks
Change of mean of pulmonary artery pressure from baseline to week 12 | At baseline and 12 weeks
Change of systolic pulmonary artery pressure from baseline to week 12 | At baseline and 12 weeks
Change of diastolic pulmonary artery pressure from baseline to week 12 | At baseline and 12 weeks
Change in Mean right atrial pressure (RAPm) | At baseline and 12 weeks
Change in Pulmonary capillary wedge pressure (PCWP) | At baseline and 12 weeks
Change in Cardiac output (CO) | At baseline and 12 weeks
Change in Mean arterial pressure (MAP) | At baseline and 12 weeks
Change Mixed venous oxygen saturation (SVO2) | At baseline and 12 weeks
Change in Systemic vascular resistance (SVR) | At baseline and 12 weeks
Change in Systemic vascular resistance index (SVRI) | At baseline and 12 weeks
Change in Cardiac index | At baseline and 12 weeks
Change in 6-minute walking test (6MWT) | At baseline, 12 weeks and 52 weeks
Change in Borg CR 10 Score | At baseline, 12 weeks and 52 weeks
Change in New York Heart Association/ World Health Organization (NYHA/WHO) class | At baseline, 12 weeks, 52 weeks and over 52 weeks
Change in N-terminal pro-B-type natriuretic peptide (NT-ProBNP) | At baseline, 12 weeks and 52 weeks
Quality of life assessed by EQ-5D and Living with Pulmonary Hypertension (LPH) questionnaires | At baseline, 12 weeks and 52 weeks
Time to clinical worsening during the study | At baseline, 12 weeks, 52 weeks and over 52 weeks
Mortality during the study | At baseline, 12 weeks, 52 weeks and over 52 weeks
Need for transplantation during the study | At baseline, 12 weeks, 52 weeks and over 52 weeks
AUC from time start of inhalation to the last data point AUC(0-tlast) | Up to 12 weeks
AUC divided by dose per kg body weight (AUCnorm) | Up to 12 weeks
AUC divided by dose (μg) (AUC/D) | Up to 12 weeks
Maximum drug concentration in plasma after start of inhalation divided by dose (μg) per kg body weight (Cmax,norm) | Up to 12 weeks
Maximum drug concentration in plasma after start of inhalation divided by dose (μg) (Cmax/D) | Up to 12 weeks
Time to reach maximum drug concentration in plasma after start of inhalation (tmax ) | Up to 12 weeks
Half-life associated with the terminal slope (t1/2) | Up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (16):
- Japan (16):
  - Nagoya, Aichi-ken
  - Kurume, Fukuoka
  - Asahikwa, Hokkaido
  - Kobe, Hyōgo
  - Kawasaki, Kanagawa
  - Sendai, Miyagi
  - Tomigusuku, Okinawa
  - Bunkyo-ku, Tokyo
  - Chuoku, Tokyo
  - Mitaka, Tokyo
  - Ōta-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Tanabe, Wakayama
  - Ube, Yamaguchi
  - Chiba
  - Tokushima

REFERENCES:
- [Result] Saji T, Myoishi M, Sugimura K, Tahara N, Takeda Y, Fukuda K, Olschewski H, Matsuda Y, Nikkho S, Satoh T. Efficacy and Safety of Inhaled Iloprost in Japanese Patients With Pulmonary Arterial Hypertension - Insights From the IBUKI and AIR Studies. Circ J. 2016;80(4):835-42. doi: 10.1253/circj.CJ-16-0097. Epub 2016 Mar 18. PMID 27001191